CLINICAL TRIAL: NCT04871269
Title: The Effect of Dronabinol on the Acquisition and Consolidation of Trauma-Associated Memories
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Stefan Roepke, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: DroMemo
Record Dates: First submitted 2021-05-03; First posted 2021-05-04 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Intrusive Memories
MeSH Terms: interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Drug: Dronabinol before the trauma film paradigm (Experimental)
  Interventions: Drug: Dronabinol; Drug: Placebo
- Drug: Dronabinol after the trauma film paradigm (Experimental)
  Interventions: Drug: Dronabinol; Drug: Placebo
- Placebo before and after the trauma film paradigm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — Dronabinol
  Arms: Drug: Dronabinol after the trauma film paradigm; Drug: Dronabinol before the trauma film paradigm
Drug: Placebo — Placebo

SUMMARY:
The aim of the current project is to investigate the impact of an activation of the cannabinoid system with an exogenous cannabinoid dronabinol (delta-9-tetrahydrocannabinol) on the formation of intrusive memories after analog trauma.

A well-established stress-film paradigm will be used to induce intrusive symptoms in healthy participants. In a double-blind placebo-controlled study, the impact of exogenous dronabinol on intrusive symptoms during exposure to a trauma film will be examined. The primary hypothesis is that exogenous oral dronabinol will decrease the number of intrusive memories recorded in the four days following experimental trauma compared with placebo controls.

This project will contribute to the current understanding of intrusive memory formation in PTSD and may guide the development of future pharmacological preventions.

DETAILED DESCRIPTION:
Recent data suggest that the cannabinoid-system is involved in stress regulation and posttraumatic stress disorder (PTSD) after traumatic events. In own of our own studies, we found reduced concentrations of the endocannabinoid arachidonylethanolamide (AEA) in BPD patients compared to healthy women (see Fig 1a). Furthermore, we found a correlation between hair concentrations of AEA and cortisol (p = .06; Fig 1b).

Low endocannabinoid signaling has been found in PTSD patients and might even present a precondition to develop PTSD after trauma. In consequence, increased endocannabinoid signaling during acquisition and consolidation of traumatic events might be a promising approach to prevent the development of PTSD. The aim of the current project is to investigate the impact of an activation of the cannabinoid system with an exogenous cannabinoid dronabinol (delta-9-tetrahydrocannabinol) on the formation of intrusive memories after analog trauma.

A well-established stress-film paradigm will be used to induce intrusive symptoms in healthy participants. In a double-blind placebo-controlled study, the impact of exogenous dronabinol on intrusive symptoms during exposure to a trauma film will be examined. The primary hypothesis is that exogenous oral dronabinol will decrease the number of intrusive memories recorded in the four days following experimental trauma compared with placebo controls.

This project will contribute to the current understanding of intrusive memory formation in PTSD and may guide the development of future pharmacological preventions.

ELIGIBILITY:
Inclusion Criteria:

* healthy female volunteers
* German on a native level

Exclusion Criteria:

* former or present disorder according to the Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5)
* any physical illnesses
* any medication intake (except oral contraceptive)
* history of traumatic experience, e.g. history of sexual abuse or rape
* pregnancy or lactation period
* follicular phase of menstrual cycle for all women not using oral contraceptives

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 291 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-08-28 (Estimated)

PRIMARY OUTCOMES:
Change of Intrusive Memories in the following four days after the intervention | four consecutive days
  Influence of dronabinol on the development of intrusive memories measured with an intrusion diary

SECONDARY OUTCOMES:
Noradrenergic System (measured with salivary alpha-amylase - u/ml) | Day 1
  Influence of dronabinol on the noradrenergic system measured with salivary alpha-amylase
Hypothalamic-pituitary-adrenal (HPA) axis (measured with salivary cortisol - nmol/L) | Time Frame: Day 1
  Influence of dronabinol on the HPA-axis measured with salivary cortisol
Polygenic Risk Score Influence of polygenic risk score on development of intrusive memories | Day 1
  Influence of polygenic risk score on development of intrusive memories

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Röpke, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany; Katja Wingenfeld, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Steglitz, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided